CLINICAL TRIAL: NCT03121313
Title: A Phase II Study of Maintenance Tegafur-uracil in Patients With Squamous Cell Carcinoma of Oral Cavity With Extracapsular Spreading of Lymph Nodes
Brief Title: Maintenance Tegafur-uracil in Resected Oral Cavity Cancer With ECS+
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103-0621A3
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2018-09

CONDITIONS: Squamous Cell Carcinoma of Oral Cavity
Keywords: Tegafur-uracil; distant metastasis; oral cavity cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms | interventions — Tegafur

STUDY DESIGN:
Intervention Model Description: Patients with resected squamous cell carcinoma of oral cavity harboring extracapsular spreading of lymph node s/p adjuvant chemoradiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maintenance (Experimental): Eligible patient will be given maintenance tegafur-uracil for one year.
  Dose of tegafur-uracil will be based on patient's body surface area (BSA):
  * BSA < 1.5 m2: tegafur-uracil 300 mg/day (1 capsule three times a day)
  * BSA ≥ 1.5 m2: tegafur-uracil 400 mg/day (2 capsules twice a day) Tegafur-uracil will be started after patient has complete the adjuvant radiotherapy and been enrolled into the study.
  Interventions: Drug: tegafur-uracil

INTERVENTIONS:
Drug: tegafur-uracil
  Other Names: UFUR

SUMMARY:
Primary Objective:

To determine the 2-year distant failure rate of maintenance tegafur-uracil in patients with squamous cell carcinoma of oral cavity with extracapsular spreading of lymph nodes.

Secondary Objectives:

* To determine the 2-year locoregional failure rate.
* To evaluate the 2-year overall survival (OS) rate.
* To evaluate the 2-year progression-free survival (PFS) rate.
* To assess the safety profiles.

DETAILED DESCRIPTION:
The primary endpoint will be 2-years distant failure rate which will be estimated by Kaplan-Meier method with two-sided 95% confidence interval.

The secondary endpoints are described as follows:

* 2-year locoregional failure rate, 2-year PFS rate and 2-year OS rate will be estimated by Kaplan-Meier method with two-sided 95% confidence interval.
* Safety profile: adverse events will be summarized by CTCAE. Safety parameters will only be analyzed on the safety analysis set and be presented in frequency tabulation.

Determination of sample size:

The estimated 2-year distant failure rate for squamous cell carcinoma of oral cavity with extracapsular spreading of lymph nodes is 26%. The 2-year distant failure rate of maintenance treatment with tegafur-uracil in this study is expected to be 13%. Using One Proportional Test with one-sided alpha 0.05 and power 80%, the sample size of 56 subjects will test an effect size of 13% (i.e. 26% vs.13%). With expected dropout rate of 20%, the sample size would be 68 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically confirmed squamous cell carcinoma with primary site in the oral cavity.
* Patient must have no distant metastasis in the pre-adjuvant radiotherapy evaluation.
* Patient must have received surgical treatment with pathologically documented extracapsular spreading of lymph node.
* Patient must have no CTCAE 4.0 grading≧2 acute adverse events from previous definite treatment at enrollment.
* Patient must can be enrolled within 1 to 3 months after definite treatment.
* Age between 20 and 70 years old;
* Patient must have ECOG performance status score 0 or 1;
* Patient must have adequate hematopoietic function which is defined as below:

  1. white blood cell (WBC) ≥ 4,000/mm3;
  2. platelet count ≥ 100,000/mm3;
  3. absolute neutrophil count (ANC) ≥ 1,500/mm3;
* Patients must have adequate hepatic function which is defined as below:

  1. serum bilirubin level < 1.5 mg/dl;
  2. sGOT and sGPT < 2.5 x ULN;
  3. serum creatinine level < 1.5 x ULN;
* All women of childbearing potential must have a negative serum or urine pregnancy test prior to the start of study medication;
* Patient with childbearing potential must agree to use a reliable contraceptive method during their participation in the study;
* Patient must have the ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Patient who has distant metastasis;
* Patient who has serious concomitant illness which might be aggravated by chemotherapy;
* Other malignancy within 5 years prior to study entry with exception of curative treated basal or squamous cell skin cancer or cervical carcinoma in situ.
* Female patient who is pregnant or breast feeding.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2015-02-26 (Actual); Primary Completion 2020-05-11 (Estimated); Study Completion 2020-05-11 (Estimated)

PRIMARY OUTCOMES:
the 2-year distant failure rate | 2 years
  the 2-year distant failure rate calculated from the date of surgery will be measured

SECONDARY OUTCOMES:
the 2-year locoregional failure rate. | 2 years
  the 2-year locoregional failure rate calculated from the date of surgery will be measured.
the 2-year overall survival (OS) rate | 2 years
  the 2-year overall survival rate calculated from the date of surgery will be measured
the 2-year progression-free survival (PFS) rate | 2 years
  the 2-year progression-free survival rate calculated from the date of surgery will be measured.
Incidence of Treatment-Emergent Adverse Events | 2 years
  Incidence of Treatment-Emergent Adverse Events will be measured by NCI-CTCAE version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Ming Wang, M.D., Principal Investigator — Chang Gung Medical Foundation
Locations (1):
- Chang-Gung Memorial Hospital-LinKou, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liao CT, Chang JT, Wang HM, Ng SH, Hsueh C, Lee LY, Lin CH, Chen IH, Huang SF, Cheng AJ, Yen TC. Analysis of risk factors of predictive local tumor control in oral cavity cancer. Ann Surg Oncol. 2008 Mar;15(3):915-22. doi: 10.1245/s10434-007-9761-5. Epub 2007 Dec 29. PMID 18165878
- [Background] Cooper JS, Pajak TF, Forastiere AA, Jacobs J, Campbell BH, Saxman SB, Kish JA, Kim HE, Cmelak AJ, Rotman M, Machtay M, Ensley JF, Chao KS, Schultz CJ, Lee N, Fu KK; Radiation Therapy Oncology Group 9501/Intergroup. Postoperative concurrent radiotherapy and chemotherapy for high-risk squamous-cell carcinoma of the head and neck. N Engl J Med. 2004 May 6;350(19):1937-44. doi: 10.1056/NEJMoa032646. PMID 15128893
- [Background] Lam P, Yuen AP, Ho CM, Ho WK, Wei WI. Prospective randomized study of post-operative chemotherapy with levamisole and UFT for head and neck carcinoma. Eur J Surg Oncol. 2001 Dec;27(8):750-3. doi: 10.1053/ejso.2001.1171. PMID 11735172
- [Background] Tsukuda M, Ogasawara H, Kaneko S, Komiyama S, Horiuchi M, Inuyama Y, Uemura T, Uchida M, Kamata S, Okuda M, et al. [A prospective randomized trial of adjuvant chemotherapy with UFT for head and neck carcinoma. Head and Neck UFT Study Group]. Gan To Kagaku Ryoho. 1994 Jul;21(8):1169-77. Japanese. PMID 8031158
- [Background] Bernier J, Domenge C, Ozsahin M, Matuszewska K, Lefebvre JL, Greiner RH, Giralt J, Maingon P, Rolland F, Bolla M, Cognetti F, Bourhis J, Kirkpatrick A, van Glabbeke M; European Organization for Research and Treatment of Cancer Trial 22931. Postoperative irradiation with or without concomitant chemotherapy for locally advanced head and neck cancer. N Engl J Med. 2004 May 6;350(19):1945-52. doi: 10.1056/NEJMoa032641. PMID 15128894
- [Background] Liao CT, Lee LY, Huang SF, Chen IH, Kang CJ, Lin CY, Fan KH, Wang HM, Ng SH, Yen TC. Outcome analysis of patients with oral cavity cancer and extracapsular spread in neck lymph nodes. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):930-7. doi: 10.1016/j.ijrobp.2010.07.1988. Epub 2010 Oct 8. PMID 20934267